CLINICAL TRIAL: NCT05380258
Title: The Effect of Chewing Gum and Use of Stress Balls on Perception of Labor Pain, Fear of Birth, and Duration of Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kastamonu University (Other)
Responsible Party: Principal Investigator, Şahika ŞİMŞEK ÇETİNKAYA, Dr. Şahika ŞİMŞEK ÇETİNKAYA, Kastamonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: KAEK-143-132
Record Dates: First submitted 2022-05-10; First posted 2022-05-18 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Labor Pain; Birth Satisfaction; Duration of Birth
Keywords: chewing gum,; stress ball; labor pain; satisfaction
MeSH Terms: conditions — Labor Pain; Personal Satisfaction | interventions — Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- chewing gum (Experimental): Pregnant women with 4-5 cm cervical dilatation started chewing gum as soon as their contractions came and they chewed gum for 20 minutes. and when the cervical dilation was 6-8 cm, they chewed gum again for 20 minutes.
  Interventions: Other: chewing gum
- stress ball (Experimental): Pregnant women with 4-5 cm cervical dilatation were asked to tighten the ball for 5 seconds and relax for 2 seconds within 20 minutes when their contractions came, and when the cervical opening was 6-8 cm, they were asked to tighten the ball for 5 seconds and relax for 2 seconds within 20 minutes.
  Interventions: Other: stress ball
- Control Group (No Intervention): standard care

INTERVENTIONS:
Other: stress ball — Pregnant women with 4-5 cm cervical dilatation were asked to tighten the ball for 5 seconds and relax for 2 seconds within 20 minutes when their contractions came, and when the cervical opening was 6-8 cm, they were asked to tighten the ball for 5 seconds and relax for 2 seconds within 20 minutes.
  Arms: stress ball
Other: chewing gum — Pregnant women with 4-5 cm cervical dilatation were asked to squeeze the ball for 5 seconds and loosen it for 2 seconds as soon as their contractions came and within 20 minutes, and when the cervical opening was 6-8 cm, they chewed gum again for 20 minutes.
  Arms: chewing gum

SUMMARY:
This study was conducted as a randomized controlled experimental study. This study was planned to determine the effects of chewing gum and using a stress ball on the perception of labor pain, duration of labor and birth satisfaction. The population of the study consisted of primiparous mothers who applied to the hospital. This study was planned to determine the effects of chewing gum and using a stress ball on the perception of labor pain, duration of labor and birth satisfaction. The study was carried out in two stages. In the first stage, the data were collected in the delivery room, and in the second stage, the postpartum satisfaction levels of the mothers were measured in the postpartum service. The sample number of the investigators' study was determined as 96. Visual analog scale, birth satisfaction scale and birth follow-up form were used for the data of our study.

ELIGIBILITY:
Inclusion Criteria:

* Being primiparous to be in due time
* To have spontaneous vaginal delivery
* Ability to communicate verbally be between the ages of 18-35
* Not having a risky pregnancy
* Having a single fetus in the vertex position
* Having started contractions and continuing regularly
* Being in the latent phase of action (0-4 cm dilatation)
* Not having used any analgesia or using any pain medication to reduce pain during labor

Exclusion Criteria:

* Mothers who have a cesarean section decision
* Risky Pregnant
* Multiple Pregnancies
* Multiparous pregnant women

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2021-06-05 (Actual); Study Completion 2022-06-05 (Actual)

PRIMARY OUTCOMES:
labor pain | Visual Analog scale I for labor pain was applied in 0-3 cm , Visual Analog Scale II in 4-5 cm and Visual Analog Scale III was applied in 6-8 cm cervical dilatation. The study continues through study completion, an average of 1 year
Duration of labor | A birth follow-up form was used from the beginning of cervical dilatation to delivery.
birth satisfaction | satisfaction form used postpartum at the 4th hour

CONTACTS AND LOCATIONS:
Locations (1):
- Şahika Şimşek Çetinkaya, Merkez, Kastamonu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No